CLINICAL TRIAL: NCT02662803
Title: Clinical, Neurophysiological and Neuroendocrine Effects of Aerobe Exercise in Generalized Anxiety Disorder (GAD)
Acronym: GAD_exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Jens Plag, physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA1/217/15
Record Dates: First submitted 2016-01-11; First posted 2016-01-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Generalized Anxiety Disorder (GAD)
Keywords: Generalized Anxiety Disorder; GAD; physical exercise; aerobe exercise; mental disorder; high-intensive aerobe exercise
MeSH Terms: conditions — Generalized Anxiety Disorder; Motor Activity; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- high-intensive aerobe exercise (Experimental): Aerobe bicycle ergometer training within 77-95% of maximum oxygen consumption; duration of each training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Interventions: Other: high-intensive aerobe exercise
- low-intensive aerobe exercise (Placebo Comparator): Aerobe training below 70% of maximum oxygen consumption (including light stretching and simple exercises adapted from yoga figures); duration of training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Interventions: Other: low-intensive aerobe exercise

INTERVENTIONS:
Other: high-intensive aerobe exercise — Aerobe bicycle ergometer training within 77-95% of maximum oxygen consumption; duration of each training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Arms: high-intensive aerobe exercise
Other: low-intensive aerobe exercise — Aerobe training below 70% of maximum oxygen consumption (including light stretching and simple exercises adapted from yoga figures); duration of training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Arms: low-intensive aerobe exercise

SUMMARY:
This study investigate the effect of high-intense aerobe exercise training (HIT) on clinical and physiological parameters (anxiety, somatisation, cortisol, alpha amylase, "mismatch negativity", loudness dependence auditory evoked potentials) in patients with generalized anxiety disorder (GAD). Half of patients will receive HIT, while the other half will receive aerobe exercise of low intensity.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a prevalent psychiatric condition and characterized by worrying of several topics of the daily life as well as stress-induced somatic symptoms (e.g. headache or musculoskeletal pain). Disturbed monoaminergic neurotransmission, changes in central information processing and altered levels of stress markers were reported as to be biological correlates of GAD or other stress-related disorders. Cognitive behavioral therapy is the first-line treatment in GAD, but it seems to be less effective than in other anxiety disorders. There is, however, some evidence for an anxiolytic activity of aerobe exercise. In this context, different forms of aerobe training were found to be associated with significant reduction of clinical symptoms in panic disorder, agoraphobia or social phobia as well as a normalisation of some of its pathophysiological markers.

In this study, 20 patients with GAD will receive a high-intensive aerobe training (HIT, 6 HIT-sessions of 20 minutes within a period of 12 days). Additionally, 20 GAD-patients will undergo a less intense aerobe training matched regarding frequency and duration of sessions. Prior to the first training session, after completing the training (day 12) and 30 days after baseline, symptoms of anxiety and somatisation will assessed by using established questionnaires. Moreover, saliva samples and electroencephalogram (EEG) will performed at the same times of assessment in order to evaluating changes of cortisol, alpha amylase, "mismatch negativity" and loudness dependence auditory evoked potentials.

We hypothesize, that GAD-patients which undergo HIT, will show a stronger and more sustained improvement of both, clinical symptoms and formally altered electrophysiological and endocrinological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Generalized Anxiety Disorder (GAD) according to the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Appropriate abilities to communicate and to complete the questionnaires
* Written informed consent
* Possibility of regular attendance at the training sessions

Exclusion Criteria:

* Other severe mental conditions than GAD (e.g. schizophrenia, severe depressive episode, addiction)
* Acute suicidality
* Epilepsy or other disorders of the central nervous system (e.g. tumor, encephalitis)
* Contraindications to aerobe exercise training
* Cardiovascular diseases
* Start or modification of an anxiolytic pharmacotherapy within the last four weeks
* Current psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in Penn State Worry Questionnaire (PSWQ, german version) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  PSWQ is a questionnaire for detecting the severity of GAD

SECONDARY OUTCOMES:
Change in Screening für somatoforme Störungen (SOMS) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  SOMS is a questionnaire for detecting the severity of somatisation
Change in Penn State Worry Questionnaire-past week (PSWQ-PW, german version) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  PSWQ-PW is a questionnaire for detecting changes in GAD-severity
Change in Screening für somatoforme Störungen - 7 Tage (SOMS-7T) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  SOMS-7T is a questionnaire for detecting changes in somatisation
Change in Hamilton Anxiety Rating Scale (HAM-A, german version) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  HAM-A is a questionnaire for detecting the severity and changes of anxiety
Change in Anxiety Control Questionnaire (ACQ, german version) | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  ACQ is a questionnaire for evaluating the ability to control anxiety
Change in saliva cortisol | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  Cortisol is an established marker of the psychophysiological stress response
Change in saliva alpha amylase | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  Alpha amylase is an established marker of the psychophysiological stress response
Change in mismatch negativity | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  Mismatch negativity is an established correlate of the central information processing
Change in loudness dependence auditory evoked potentials | From baseline to post therapy (+12 days) and from baseline to follow-up (+30 days)
  Loudness dependence auditory evoked potentials are established correlates of the central serotonergic transmission

CONTACTS AND LOCATIONS:
Overall Officials: Plag JP Plag, Dr., Study Chair — Department of Psychiatry and Psychotherapy, Charité - Universitätsmedizin Berlin, Campus Mitte
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité - Universitätsmedizin Berlin, Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaudlitz K, Plag J, Dimeo F, Strohle A. Aerobic exercise training facilitates the effectiveness of cognitive behavioral therapy in panic disorder. Depress Anxiety. 2015 Mar;32(3):221-8. doi: 10.1002/da.22337. Epub 2014 Dec 17. PMID 25515221
- [Background] Ghisolfi ES, Heldt E, Zanardo AP, Strimitzer IM Jr, Prokopiuk AS, Becker J, Cordioli AV, Manfro GG, Lara DR. P50 sensory gating in panic disorder. J Psychiatr Res. 2006 Sep;40(6):535-40. doi: 10.1016/j.jpsychires.2006.02.006. Epub 2006 Apr 17. PMID 16616936
- [Background] Hegerl U, Juckel G. Intensity dependence of auditory evoked potentials as an indicator of central serotonergic neurotransmission: a new hypothesis. Biol Psychiatry. 1993 Feb 1;33(3):173-87. doi: 10.1016/0006-3223(93)90137-3. PMID 8383545
- [Background] Clark CR, McFarlane AC, Weber DL, Battersby M. Enlarged frontal P300 to stimulus change in panic disorder. Biol Psychiatry. 1996 May 15;39(10):845-56. doi: 10.1016/0006-3223(95)00288-x. PMID 9172705
- [Background] Naatanen R. The mismatch negativity: a powerful tool for cognitive neuroscience. Ear Hear. 1995 Feb;16(1):6-18. PMID 7774770
- [Background] Plag J, Gaudlitz K, Schumacher S, Dimeo F, Bobbert T, Kirschbaum C, Strohle A. Effect of combined cognitive-behavioural therapy and endurance training on cortisol and salivary alpha-amylase in panic disorder. J Psychiatr Res. 2014 Nov;58:12-9. doi: 10.1016/j.jpsychires.2014.07.008. Epub 2014 Jul 21. PMID 25085607
- [Background] Schumacher S, Kirschbaum C, Fydrich T, Strohle A. Is salivary alpha-amylase an indicator of autonomic nervous system dysregulations in mental disorders?--a review of preliminary findings and the interactions with cortisol. Psychoneuroendocrinology. 2013 Jun;38(6):729-43. doi: 10.1016/j.psyneuen.2013.02.003. Epub 2013 Mar 5. PMID 23481259
- [Background] Burgomaster KA, Hughes SC, Heigenhauser GJ, Bradwell SN, Gibala MJ. Six sessions of sprint interval training increases muscle oxidative potential and cycle endurance capacity in humans. J Appl Physiol (1985). 2005 Jun;98(6):1985-90. doi: 10.1152/japplphysiol.01095.2004. Epub 2005 Feb 10. PMID 15705728
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Stober J, Bittencourt J. Weekly assessment of worry: an adaptation of the Penn State Worry Questionnaire for monitoring changes during treatment. Behav Res Ther. 1998 Jun;36(6):645-56. doi: 10.1016/s0005-7967(98)00031-x. PMID 9648338
- [Background] Maier W, Buller R, Philipp M, Heuser I. The Hamilton Anxiety Scale: reliability, validity and sensitivity to change in anxiety and depressive disorders. J Affect Disord. 1988 Jan-Feb;14(1):61-8. doi: 10.1016/0165-0327(88)90072-9. PMID 2963053
- [Background] Plag J, Schumacher S, Strohle A. [Generalized anxiety disorder]. Nervenarzt. 2014 Sep;85(9):1185-94. doi: 10.1007/s00115-014-4121-8. German. PMID 25119343
- [Background] Jayakody K, Gunadasa S, Hosker C. Exercise for anxiety disorders: systematic review. Br J Sports Med. 2014 Feb;48(3):187-96. doi: 10.1136/bjsports-2012-091287. Epub 2013 Jan 7. PMID 23299048